CLINICAL TRIAL: NCT07306104
Title: The Effect of Long-term Treatment of Parkinson's Disease With T-PEMF
Brief Title: The Effect of Long-term Daily Stimulation of the Brain With Pulsed Electromagnetic Fields on Parkinsons Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Bente & Erik Schøller Larsens Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDURio #12.562; 2501906 (Other: The Danish Medical Research Ethics Committees)
Record Dates: First submitted 2025-11-21; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: T-PEMF
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking only applies to the intervention groups. The control group and reference group are Open Label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention group 1: Full T-PEMF (Experimental): Persons with Parkinson's disease receiving 30 min daily active T-PEMF for 12 months. The first 6 months are blinded, the last 6 months are not.
  Interventions: Device: Transcranial pulsed electromagnetic fields (T-PEMF)
- Intervention group 2: sham + T-PEMF (Sham Comparator): Persons with Parkinson's disease receiving 30 min daily sham T-PEMF for 6 months followed by 6 moths of 30 min daily active T-PEMF. The first 6 month is blinded, the last 6 months are not.
  Interventions: Device: Transcranial pulsed electromagnetic fields (T-PEMF); Device: Sham (No Treatment)
- Control group (No Intervention): Persons with Parkinson's disease receiving no experimental treatment. The group is used to monitor natural course of the disease.
- Healthy reference group (No Intervention): Health age-matched persons assessed once to obtain age-matched normal intervals of performance.

INTERVENTIONS:
Device: Transcranial pulsed electromagnetic fields (T-PEMF) — 30 min daily stimulation with transcranial pulsed electromagnetic fields (50 Hz)
  Arms: Intervention group 1: Full T-PEMF; Intervention group 2: sham + T-PEMF
Device: Sham (No Treatment) — 30 min daily the participants are using/wearing the T-PEMF device but no stimulation occurs
  Arms: Intervention group 2: sham + T-PEMF

SUMMARY:
The goal of this clinical trial is to learn to what extent daily stimulation of the brain with transcranial pulsed electromagnetic fields (T-PEMF) works to treat persons with Parkinson's Disease. The main questions it aims to answer are:

* How does 6 months of daily treatment (30 minutes/day) with T-PEMF affects neuro-mechanical and molecular biological factors compared with placebo treatment in persons with Parkinson's disease?
* How does 12 months of daily treatment (30 minutes/day) with T-PEMF affects neuro-mechanical and molecular biological factors in persons with Parkinson's disease an does 12 months of T-PEMF alters the need for medication intake?

The neuro-mechanical outcomes are compared with the "natural" progression of the disease as well as with a healthy reference group. Furthermore, it will be examined whether 12 months of T-PEMF treatment alters the need for medication intake.

Participants in the intervention group will:

* receive one 30 min treatment session daily for 12 months
* receive either T-PEMF or sham treatment for the first 6 months
* receive active T-PEMF treatment the last 6 months
* visit for tests before treatment initiation, after 6 months of treatment and after 12 months of treatment.

ELIGIBILITY:
Intervention Groups

Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease
* The participant must be able to understand, accept, and complete the planned procedures
* Parkinson's symptoms in the medicated state must correspond to Hoehn & Yahr stage 1 or 2
* Mini Mental-State Examination score > 22

Exclusion Criteria:

* Cancer in the brain, neck, or head area
* Presence of active medical implants
* Epilepsy
* Alcoholism
* Substance abuse
* Open wound on the scalp
* Severe psychopathological disorders
* Pregnancy
* Changes in pharmacological anti-Parkinson medication within the last 6 weeks prior to the start of T-PEMF treatment
* Anticoagulant treatment with Marevan, Marcoumar, Pradaxa, Eliquis, Xarelto, Lixiana, Novostan, Fragmin, or Innohep
* Neurological disease other than Parkinson's disease
* Previous stroke
* Reduced motor function caused by conditions other than Parkinson's disease

Control Group with Parkinson's Disease

Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease
* The patient must be able to understand, accept, and complete the planned procedures
* Parkinson's symptoms in the medicated state must correspond to Hoehn & Yahr stage 1 or 2
* Mini Mental-State Examination score > 22

Exclusion Criteria:

* Neurological disease other than Parkinson's disease
* Reduced motor function caused by conditions other than Parkinson's disease

Healthy Reference Group:

Inclusion Criteria:

-The patient must be able to understand, accept, and complete the planned procedures

Exclusion Criteria:

* Neurological disease
* Reduced motor function caused by condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Sit-to-stand | From enrollment to end of intervention assessed at baseline, after 6 months and after 12 months.
  Completion time of 5 repetition sit-tot-stand test at maximal speed performed on force plate.

SECONDARY OUTCOMES:
Tremor intensity | From enrollment to end of intervention assessed at baseline, after 6 months and after 12 months.
  Postural tremor intensity assessed by accelerometer
Rate of force development | From enrollment to end of intervention assessed at baseline, after 6 months and after 12 months.
  Isometric rate of force development assessed by handgrip and knee extension
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | From enrollment to end of intervention assessed at baseline, after 6 months and after 12 months.
  The MDS-UPDRS will be reported as total score (0-260, higher scores indicate greater disease severity) and motor score (part III, 0-132, higher scores indicate greater disease severity).
Cerebrospinal fluid biomarkers | From enrollment to end of intervention assessed at baseline, after 6 months and after 12 months. Assessment in the intervention groups only.
  Concentration of growth factors, cytokines and cytoskeletal proteins with special emphasis on erythropoietin (EPO), vascular endothelial growth factor (VEGF), brain-derived neutrophic factor (BDNF), glia cell derived neutrophilic factor (GDNF), Glucagon Like Peptide 1 (GLP1), interleukins and neurofilament light chain (NfL).

OTHER OUTCOMES:
EMG | From enrollment to end of intervention assessed at baseline, after 6 months and after 12 months.
  Electromyographic recordings of forearm and thigh muscles during motor assessments (sit-to-stand, isometric contractions, postural tremor assessment, handwriting). Applied for explorative analyses, thus exact outcomes are not yet specified. However, agonist drive and co-contraction ratio may be assessed.
Hand writing | From enrollment to end of intervention assessed at baseline, after 6 months and after 12 months.
  Hand writing test performed with ink pen on paper on top of tablet (digitalizing handwriting). Performed as an explorative assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sofie Bøgh Malling, Ph.d., Principal Investigator — University of Southern Denmark
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense
  - University of Southern Denmark, Odense

IPD SHARING:
Plan to Share IPD: No